CLINICAL TRIAL: NCT03031990
Title: Yoga and Infertility: The Impact of Yoga on Anxiety Reduction in Patients Undergoing in Vitro Fertilization or Elective Oocyte Freezing
Brief Title: Stress and Fertility: How to Lower Stress When Trying to Conceive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fertility Centers of Illinois (Other)
Collaborators: Pulling Down the Moon, Holistic Health (Unknown); Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15121505
Record Dates: First submitted 2017-01-04; First posted 2017-01-26 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Anxiety; Infertility, Female
Keywords: Yoga; Oocyte cryopreservation; In-vitro fertilization
MeSH Terms: conditions — Anxiety Disorders; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga intervention (Experimental): The participants who elect to include yoga as part of their infertility treatments will self select one of three groups: 1) In person yoga for fertility group; 2) Online yoga for fertility group; 3) In person discussion only group
  Interventions: Behavioral: In-person yoga for fertility group; Behavioral: Online yoga for fertility group; Behavioral: In person discussion only group
- Control (No Intervention): These are patients that have a history of IVF failure or who are undergoing elective egg freezing who elect to be included in the study but are not interested in including yoga as a part of their treatment.

INTERVENTIONS:
Behavioral: In-person yoga for fertility group — The participants in this group will complete the Yoga for Fertility class at Pulling Down the Moon: An Integrative Center for Fertility. This consists of a 30 minute discussion session followed by a 60 minute Vinyasa style yoga class one time a week for a total of 6 weeks. Participants must attend at least 5 out of the 6 sessions to be included in the analysis.
  Arms: Yoga intervention
Behavioral: Online yoga for fertility group — The participants in this group will complete an online webinar of the Yoga for Fertility class and engage in a home yoga practice with the Pulling Down the Moon Yoga DVD. This will occur one time a week for a total of 6 weeks. Participants must complete at least 5 out of the 6 sessions to be included in the analysis.
  Arms: Yoga intervention
Behavioral: In person discussion only group — The participants in this group will attend an in-person 30 minute discussion session at Pulling Down the Moon. This will occur one time a week for a total of 6 weeks. Participants must complete at least 5 out of the 6 sessions to be included in the analysis.
  Arms: Yoga intervention

SUMMARY:
Psychological stress and its sources differ among the population and can be reduced in various ways. The practice of yoga has been shown to be an effective stress reducing agent. IVF processes have also been shown to increase stress levels, particularly in patients with multiple failed IVF cycles. Less is known about stress levels in patients undergoing elective egg freezing for fertility preservation. The investigators demonstrated in a pilot project that yoga postures with a yoga focused discussion session decreases stress in infertility patients compared to controls. The goal of this study is to further explore the capability of yoga practice to reduce stress in a specific subset of infertility patients, those with a history of at least one failed IVF cycle and those undergoing elective oocyte cryopreservation. Additionally, the investigators are aiming to understand which aspect of the intervention (discussion vs. yoga) had the most impact and whether route of administration of the intervention (in person vs online) effects results.

DETAILED DESCRIPTION:
Although stress is likely not a cause of infertility, research has shown negative effects of psychological stress on in vitro fertilization (IVF) outcomes. IVF processes have also been shown to increase stress in infertility patients. Patients that have had failed at IVF cycles are noted to have more stress. The practice of elective egg freezing is relatively new and little is known on the psychological wellbeing of these patients as they start ovarian stimulation for egg freezing. The practice of yoga has been shown to be an effective stress reducing agent. The investigators demonstrated in a pilot project that yoga postures coupled with a yoga focused discussion session decreases stress in infertility patients compared to controls. Therefore, the purpose of this study is to further explore this relationship and determine which aspect of the intervention had the most impact.

Participants will include women with a history of at least one IVF failure or women undergoing fertility preservation for elective egg freezing. The participants who elect to include yoga as part of their infertility treatments will self select one of three treatment groups: 1) In person yoga + discussion; 2) online yoga + discussion; 3) In person discussion only. The investigators will also recruit non-yoga participators as a control group.

The yoga participants and controls will be asked to fill out two questionnaires: The State-Trait Anxiety Inventory (STAI) and the Fertility Problem Inventory (FPI). STAI is a widely used measure of trait anxiety (a person's disposition towards being anxious over time) and state anxiety (how anxious a person feels at the present time). It is a 40-question survey that uses a 4-point Likert scale per question. A score of 20 corresponds to low anxiety and a score of 80 corresponds to high anxiety. It has been shown that higher anxiety scores exist in the infertility population. Mean STAI scores in the infertility population range between 30-50. The FPI is used as another tool for assessing a person's state anxiety and has been found to better discriminate between general stress and infertility-related stress. Participants will complete these at the beginning of participation and then again six weeks later. The design of the study will include a pre-test and post-test analysis.

The primary outcome is to determine whether stress reduction is greater in those women that participate in the yoga postures and discussion group when compared to those in the discussion only group or controls. The secondary hypothesis is that reduction in stress will be equivalent between online and in-person participators. Additional outcomes include an assessment of whether age or other demographic factors influence baseline stress levels or reduction in stress. The investigators also plan to examine whether the yoga participation has any influence on ovarian stimulation or pregnancy outcomes. Therefore, baseline patient demographic characteristics, clinical outcomes regarding ovarian stimulation as well as future pregnancy outcomes will also be collected.

The investigators plan to recruit at least 150 participants who are currently undergoing in-vitro fertilization (IVF) at Fertility Centers of Illinois (FCI) and 150 patients undergoing elective egg freezing for fertility preservation at FCI. Those 150 patients will then be further subdivided into one of the three treatment groups mentioned above or the control group.

Before starting the study, the participants interested in a treatment group involving yoga postures will be evaluated including a review of medical history and an assessment of ability to perform basic, gentle yoga without injury. All interventions will occur once weekly for a total of six weeks. The participant will be expected to participate in at least five of the six sessions in order to complete the study. If the participant is in the in person yoga + discussion group, she will complete a Yoga for Fertility class Pulling Down the Moon: An Integrative Center for Fertility which consists of a 30 minute discussion session followed by a 60 minute Vinyasa style yoga class. If the participant is in the online yoga + discussion group, she will attend an online webinar of the Yoga for Fertility class and engage in a home yoga practice with the Pulling Down the Moon Yoga DVD. If the participant is in the discussion only group, she will attend an in-person 30 minute discussion session at Pulling Down the Moon.

The investigators will be using paired t-tests to compare mean pre-test and post-test scores between groups and logistic regressions to evaluate the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of one prior IVF failure and planning to undergo a subsequent IVF cycle at the Fertility Centers of Illinois (FCI) OR
* Patients undergoing elective egg freezing for fertility preservation at FCI
* Deemed medically able to perform basic, gentle yoga without injury

Exclusion Criteria:

* Other medical problems that preclude yoga participation (though may be eligible for control group participation)

Ages: 24 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Stress levels pre and post intervention between groups using STAI | 6 weeks
  Will evaluate by comparing mean pre and post test scores for the State-Trait Anxiety Inventory (STAI) between groups to determine which treatment option produced highest reductions in anxiety. The STAI is a 40 question questionnaire scored on a point scale from 20-80.
Stress levels pre and post intervention between groups using FPI | 6 weeks
  Will evaluate by comparing mean pre and post test scores for the The Fertility Problem Inventory (FPI) between groups to determine which treatment option produced highest reductions in anxiety. The FPI is a 46 question questionnaire scored by generating a composite score from five sub scale scores.

SECONDARY OUTCOMES:
Difference between mean pre and post STAI test scores between in person and online yoga for fertility programs | 6 weeks
  Will compare mean pre and post test scores on STAI between the in person and online yoga for fertility groups to determine whether the reduction in stress was greater in one versus the other.
Difference between mean pre and post FPI test scores between in person and online yoga for fertility programs | 6 weeks
  Will compare mean pre and post test scores on FPI between the in person and online yoga for fertility groups to determine whether the reduction in stress was greater in one versus the other.
Influence of ethnicity on baseline stress levels and reduction in stress using the STAI | 6 weeks
  Will compare mean pre and post test scores on STAI between various ethnic groups (1=American Indian/Native American, 2=Arab, 3=Asian/Pacific Islander, 4=Black/African American, 5=Caucasian/White, 6=Hispanic/Latino, 7=Multiracial, 8=Other, 9=Prefer not to answer).
Influence of ethnicity on baseline stress levels and reduction in stress using FPI | 6 weeks
  Will compare mean pre and post test scores on FPI between various ethnic groups (1=American Indian/Native American, 2=Arab, 3=Asian/Pacific Islander, 4=Black/African American, 5=Caucasian/White, 6=Hispanic/Latino, 7=Multiracial, 8=Other, 9=Prefer not to answer).
Influence of age on baseline stress levels and reduction in stress using STAI | 6 weeks
  Will compare mean pre and post test scores on STAI across ages (ranging 24-42).
Influence of age on baseline stress levels and reduction in stress using FPI | 6 weeks
  Will compare mean pre and post test scores on FPI across ages (ranging 24-42).
Influence of number of previous IVF failures on baseline stress levels and reductions in stress using STAI | 6 weeks
  Will compare mean pre and post test scores on STAI between participants when grouped based on the number of prior IVF failures.
Influence of number of previous IVF failures on baseline stress levels and reductions in stress using FPI | 6 weeks
  Will compare mean pre and post test scores on FPI between participants when grouped based on the number of prior IVF failures.
Influence of yoga participation on number of days required for ovarian stimulation | 6 weeks
  Will compare the above outcome between treatment groups as well as to the control group
Influence of yoga participation on number of oocytes obtained | 6 weeks
  Will compare the above outcome between treatment groups as well as to the control group
Influence of yoga participation on number of mature (M2) oocytes | 6 weeks
  Will compare the above outcome between treatment groups as well as to the control group
Influence of yoga participation on fertilization rate | 6 weeks
  Will compare the above outcome between treatment groups as well as to the control group
Influence of yoga participation on number of high quality embryos (as evidenced by embryologists embryo grading criteria) | 6 weeks
  Will compare the above outcome between treatment groups as well as to the control group
Influence of yoga participation on rates of positive pregnancy test | 1 year
  Will follow patients who achieve pregnancy in cycle following intervention and track pregnancy outcomes to determine if there was a difference in outcomes between treatment and control groups.
Influence of yoga participation on clinical pregnancy rate | 1 year
  Will follow patients who achieve pregnancy in cycle following intervention and track pregnancy outcomes to determine if there was a difference in outcomes between treatment and control groups.
Influence of yoga participation on ongoing pregnancy/live birth rate | 1 year
  Will follow patients who achieve pregnancy in cycle following intervention and track pregnancy outcomes to determine if there was a difference in outcomes between treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hirshfeld, MD, Study Director — Fertility Centers of Illinois; Anne E Martini, DO, Principal Investigator — Rush University Medical Center; Beth Heller, MS, Study Director — Pulling Down the Moon, Holistic Health
Locations (1):
- Fertility Centers of Illinois, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jasani S, Heller B, Jasulaitis S, Davidson M, Cytron JH. Impact of a Structured Yoga Program on Anxiety in Infertility Patients: A Feasibility Study. JFIV Reprod Med Genet 4: 183, 2016.
- [Background] Domar AD, Zuttermeister PC, Friedman R. The psychological impact of infertility: a comparison with patients with other medical conditions. J Psychosom Obstet Gynaecol. 1993;14 Suppl:45-52. PMID 8142988
- [Background] Sanders KA, Bruce NW. Psychosocial stress and treatment outcome following assisted reproductive technology. Hum Reprod. 1999 Jun;14(6):1656-62. doi: 10.1093/humrep/14.6.1656. PMID 10357996
- [Background] Ebbesen SM, Zachariae R, Mehlsen MY, Thomsen D, Hojgaard A, Ottosen L, Petersen T, Ingerslev HJ. Stressful life events are associated with a poor in-vitro fertilization (IVF) outcome: a prospective study. Hum Reprod. 2009 Sep;24(9):2173-82. doi: 10.1093/humrep/dep185. Epub 2009 May 22. PMID 19465459
- [Background] Domar AD, Gross J, Rooney K, Boivin J. Exploratory randomized trial on the effect of a brief psychological intervention on emotions, quality of life, discontinuation, and pregnancy rates in in vitro fertilization patients. Fertil Steril. 2015 Aug;104(2):440-51.e7. doi: 10.1016/j.fertnstert.2015.05.009. Epub 2015 Jun 13. PMID 26072382
- [Background] Lawson AK, Klock SC, Pavone ME, Hirshfeld-Cytron J, Smith KN, Kazer RR. Prospective study of depression and anxiety in female fertility preservation and infertility patients. Fertil Steril. 2014 Nov;102(5):1377-84. doi: 10.1016/j.fertnstert.2014.07.765. Epub 2014 Aug 22. PMID 25154674
- [Background] Oron G, Allnutt E, Lackman T, Sokal-Arnon T, Holzer H, Takefman J. A prospective study using Hatha Yoga for stress reduction among women waiting for IVF treatment. Reprod Biomed Online. 2015 May;30(5):542-8. doi: 10.1016/j.rbmo.2015.01.011. Epub 2015 Feb 3. PMID 25779021
- [Background] Domar AD, Rooney KL, Wiegand B, Orav EJ, Alper MM, Berger BM, Nikolovski J. Impact of a group mind/body intervention on pregnancy rates in IVF patients. Fertil Steril. 2011 Jun;95(7):2269-73. doi: 10.1016/j.fertnstert.2011.03.046. Epub 2011 Apr 15. PMID 21496800
- [Background] Khalsa HK. Yoga: an adjunct to infertility treatment. Fertil Steril. 2003 Oct;80 Suppl 4:46-51. doi: 10.1016/s0015-0282(03)01138-5. PMID 14568288
- [Background] Galhardo A, Cunha M, Pinto-Gouveia J. Mindfulness-Based Program for Infertility: efficacy study. Fertil Steril. 2013 Oct;100(4):1059-67. doi: 10.1016/j.fertnstert.2013.05.036. Epub 2013 Jun 27. PMID 23809500
- [Background] Newham JJ, Westwood M, Aplin JD, Wittkowski A. State-trait anxiety inventory (STAI) scores during pregnancy following intervention with complementary therapies. J Affect Disord. 2012 Dec 15;142(1-3):22-30. doi: 10.1016/j.jad.2012.04.027. Epub 2012 Sep 7. PMID 22959685
- [Background] Newton CR, Sherrard W, Glavac I. The Fertility Problem Inventory: measuring perceived infertility-related stress. Fertil Steril. 1999 Jul;72(1):54-62. doi: 10.1016/s0015-0282(99)00164-8. PMID 10428148